CLINICAL TRIAL: NCT04996979
Title: Evaluation of the PENG Block vs Placebo for Preoperative Pain Control in Hip Fractures in the Elderly - a Double-blinded Randomised Controlled Trial
Brief Title: Patients With Acute Hip Fractures Will Receive Either the PENG Block or no Block Respectively.
Acronym: PENGBlock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2021-05-10; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Hip Fractures
Keywords: Hip fractures, elderly, pain
MeSH Terms: conditions — Hip Fractures; Pain | interventions — Ropivacaine; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient, nurses and CRC will be blinded. Rest of study team is not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Only standard care
  Interventions: Drug: Placebo
- Intervention group (Experimental): The PENG block was performed for intervention group with local anaesthetic solution composed of 20 ml of ropivacaine 0.5%.
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.5% Injectable Solution — Local anaesthetic solution composed of ropivacaine 0.5%(intervention group)
  Arms: Intervention group
Drug: Placebo — Standard care
  Other Names: Standard care
  Arms: Control

SUMMARY:
Hip fracture pain is often severe and traditionally managed by systemic opioids which have increased risk of side effects in frail elderly patients. Inadequately controlled pain may lead to delirium which increases mortality and morbidity. The overall aim of this RCT is to investigate the potential for improved pain relief accomplished by the addition of the PENG block to current standard practice of pre-operative analgesia (systemic morphine), compared to the control group, which involves no block (operator will still go through the motion as if performing a block) plus standard pre-operative analgesia.

The investigator hypothesize that the addition of a single shot PENG block at the side of hip fracture in addition to traditional systemic morphine provides good preoperative pain relief on movement and reduces the need for breakthrough opioid requirements. The investigator hypothesize that the interventional group dynamic pain score assessed at 30 minutes after the block compared to control group dynamic pain score at 30 minutes after the "block" will be at least a 3 point difference between the 2 groups .

DETAILED DESCRIPTION:
Specific Aim1: To determine difference in pain scores on movement (dynamic pain scores) in patients who receive the PENG block in the intervention group compared to no block in the control group at 30 minutes after performance of the block.

Specific Aim2: To determine if there is any difference in pain at rest between the intervention group and the control group, and if so, the magnitude of the difference in pain scores.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 years old and above
2. Provided consent for the study
3. Patients with solitary hip fracture (no other fracture) - intracapsular neck of femur fracture, intertrochanteric fracture
4. Either awaiting hip fracture surgery or no plans for hip fracture surgery within the next 24 hours

Exclusion Criteria:

1. Patients with cognitive impairment or inability to give consent, or refusal to give consent
2. Multiple fracture cases
3. Peri-prosthetic fractures and revisions
4. Subclinical vertebral fractures
5. Hip fractures due to major accidents such as road traffic accidents, fall from height or more than 2 meters
6. Multiple trauma
7. Pathological fractures secondary to metastases
8. Patients with contraindications to block performance

   * Coagulopathy as demonstrated by PT/PTT/INR
   * On antiplatelets or anticoagulation
   * Infection/ compromised skin integrity at site of block performance
   * Allergy to local anaesthetics and opioids

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Dynamic pain scores (Numerical pain score (NRS) at 15 degrees leg lift) | 30 minutes after receiving intervention
  The difference in dynamic pain scores (NRS at 15 degrees leg lift) at 30 minutes post block performance in the intervention group vs the control group. Assessment of the dynamic pain score is done prior to discharge from recovery at SGH Pain Management Centre.

SECONDARY OUTCOMES:
Pain scores (NRS) at rest (static pain) and on movement (dynamic pain) | Up to 24 hours from performance of block
  It is measured at Baseline, Immediately after performance of block, 30 minutes after the lock in recovery At 60 minutes, 180 minutes and 24 hours post block in the ward
Pain scores collected to estimate the onset and duration of block Pain scores to estimate the onset and duration of block | Up to 24 hours from performance of block
  Taking the recorded time taken for the pain relieve to estimate onset time using models
Total opioid use over 24 hours as a surrogate measure | Up to 24 hours from performance of block
  Using the data recorded for :
  Oral morphine use Intravenous morphine use for patients on PCA Doses of opioid use will be converted to morphine milligram equivalent daily dose (MEDD) for standardized comparison.

CONTACTS AND LOCATIONS:
Locations (1):
- Pain Management Center Sinagpore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tay E. Hip fractures in the elderly: operative versus nonoperative management. Singapore Med J. 2016 Apr;57(4):178-81. doi: 10.11622/smedj.2016071. PMID 27075376
- [Result] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Derived] Lin X, Liu CW, Goh QY, Sim EY, Chan SKT, Lim ZW, Chan DXH. Pericapsular nerve group (PENG) block for early pain management of elderly patients with hip fracture: a single-center double-blind randomized controlled trial. Reg Anesth Pain Med. 2023 Nov;48(11):535-539. doi: 10.1136/rapm-2022-104117. Epub 2023 Apr 13. PMID 37055189
- See also: Anaesthetic management of patients with hip fractures: an update — https://doi.org/10.1093/bjaceaccp/mkt006